CLINICAL TRIAL: NCT03276702
Title: A Protocol for Prospectively Collecting Fresh Tumor Tissue in Children and Adolescents With Recurrent or Progressive Solid Malignancies
Brief Title: Tumor Rebiopsy in Children and Adolescents With Recurrent or Progressive Solid Malignancies
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REBIOP
Record Dates: First submitted 2017-09-07; First posted 2017-09-08 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Tumor, Solid
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be extracted from the patient's peripheral blood and tumor samples and RNA will be extracted from the tumor sample and whole genome sequencing (WGS), whole exome sequencing (WES) and transcriptome sequencing (RNA-Seq) will be performed on Illumina Next Generation Sequencers. Both somatic and germline variants (single nucleotide variants, structural variants, insertions/deletions, and copy number variants) will be identified using a bioinformatics pipeline developed and validated at SJCRH. Separate reports will be generated for the somatic lesions and germline lesions. In the event that there is not enough fresh tissue to perform WGS, WES and RNAseq will be performed in FFPE material if available.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: St. Jude Children's Research Hospital patients with relapsed or progressive solid tumor will be asked to complete a questionnaire on two occasions and optional re-biopsy of tumor tissue.
  Interventions: Procedure: Re-biopsy; Other: Questionnaire

INTERVENTIONS:
Procedure: Re-biopsy — For those participants who agree, a biopsy of their tumor to obtain tissue for genetic analysis will be done at the time of relapse or disease progression.
  Other Names: Tumor tissue biopsy
Other: Questionnaire — Parents or patients will be asked to complete a questionnaire to assess the impact and perception of an optional/research only biopsy. A second questionnaire will be administered approximately 4-8 weeks after biopsy to assess decisional regret.
  Other Names: Assessment

SUMMARY:
It has been shown that the genomic landscape of tumors can dramatically change at the time of disease progression. This suggests that therapies aimed at treating the tumor at diagnosis may not be relevant at the time of relapse. Obtaining fresh tissue at the time of relapse could facilitate the identification of potential targets that have developed through mutational evolution of the primary tumor and would provide an unprecedented opportunity to expand the library of patient derived xenografts (PDX) that are available for comprehensive preclinical testing in the setting of relapsed disease.

The purpose of this observational study is to prospectively collect fresh tumor tissue from pediatric patients with solid tumors who have recurrent or progressive disease and submit this tissue for comprehensive genomic analysis using clinically available CLIA-certified platforms that include WGS, WES and RNAseq, and to assess the reasons for a patient and/or a parent for making a decision to proceed with or refuse a re-biopsy procedure in the presence of a recurrent or progressive solid tumor. The data obtained will be used to develop new novel therapies that incorporate new pharmacological agents in pediatric solid tumors.

PRIMARY OBJECTIVES:

* To prospectively collect fresh tumor tissue from pediatric patients with solid tumors who have recurrent or progressive disease and submit this tissue for comprehensive genomic analysis.
* To assess the reasons a patient and/or a parent make the decision to proceed with or refuse a re-biopsy procedure in the presence of a recurrent or progressive solid tumor.

SECONDARY OBJECTIVES:

* To estimate refusal and acceptance rates for re-biopsy and the parental/patient attitudes towards a re-biopsy.
* To estimate the incidence of complications associated with biopsy.
* To estimate the percentage of procedures that fail to obtain adequate tissue for genomic analysis.

DETAILED DESCRIPTION:
This is a prospective, non-therapeutic study with two components: biopsy of tumor for genomic studies and prospective assessment of parental factors related to participation. All patients at St. Jude Children's Research Hospital (SJCRH) who meet the eligibility criteria will be approached for study participation. The re-biopsy is not mandatory and will only be performed after the patient and family have consented. A questionnaire to assess the impact and perception of an optional/research only biopsy will be administered following the decision regarding re-biopsy. For those consenting to the re-biopsy, approximately 4-8 weeks after biopsy, the family and patient will be asked to complete a second questionnaire to assess decisional regret.

Participants may repeat participation in this trial with subsequent relapses, provided informed consent is obtained prior to each re-biopsy procedure. For those participants who consent to repeat participation, all protocol procedures will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-21 years
* Patient has been diagnosed with a solid tumor malignancy that is recurrent or progressive and for whom there is no fresh tumor specimen available.
* Availability of gross disease amenable to biopsy.
* Karnofsky ≥ 50% for patients >16 years of age and Lansky ≥ 50 for patients ≤ 16 years of age.

Exclusion Criteria:

* Diagnosis of a non-solid tumor malignancy.
* Patient with known coagulopathy that requires replacement therapy.
* Patient with anesthesia risk that would place the patient at a higher than expected risk for complications (ASA PS4 and ASA PS5).
* Karnofsky or Lansky performance score of < 50.
* BMI for age > 95th percentile.
* Refusal or inability to provide written informed consent according to institutional guidelines.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: St. Jude Children's Research Hospital patient with a solid tumor malignancy that is progressive or recurrent.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Percent of good quality tumor samples obtained | Once at study enrollment
  Good quality of the sampled tumor is defined as greater than 50% viable tumor from which at least 2 µg DNA and 1 µg RNA can be extracted.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Pappo, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols